CLINICAL TRIAL: NCT00002412
Title: A Randomized, Double-Blind Study of MKC-442 Combined With Stavudine, Didanosine, and Hydroxyurea in HIV-Infected Patients Who Are Protease Inhibitor Experienced and Non-Nucleoside Reverse Transcriptase Inhibitor Naive
Brief Title: A Study of MKC-442 in Combination With Other Anti-HIV Drugs
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Triangle Pharmaceuticals (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: 292C; MKC-305
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1999-04

CONDITIONS: HIV Infections
Keywords: Didanosine; Drug Therapy, Combination; Stavudine; Hydroxyurea; Reverse Transcriptase Inhibitors; Anti-HIV Agents; Viral Load; MKC 442
MeSH Terms: conditions — HIV Infections | interventions — emivirine; Hydroxyurea; Stavudine; Didanosine

INTERVENTIONS:
Drug: Emivirine
Drug: Hydroxyurea
Drug: Stavudine
Drug: Didanosine

SUMMARY:
The purpose of this study is to see if it is safe and effective to give MKC-442 plus stavudine (d4T) plus didanosine (ddI) plus hydroxyurea.

DETAILED DESCRIPTION:
Patients are randomized to receive either MKC-442 or placebo, along with stavudine(d4T), didanosine(ddI), and hydroxyurea. Patients will be treated and followed for 48 weeks.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

- Based on medical history, medical condition, prior use of antiretroviral drugs, and genotypic analysis of the predominant strain of HIV-1 isolated from the plasma, administration of a combination of two or more available antiretroviral agents by prescription may be given with MKC-442.

Patient must have:

* HIV infection with HIV-1 RNA greater than or equal to 5,000 by Roche Amplicor method within 30 days of entry.
* A failed protease inhibitor-containing regimen.
* Negative serum beta human chorionic gonadotropin test within 30 days of entry.

Prior Medication:

Allowed:

* Prior nucleoside reverse transcriptase and protease inhibitors.
* Cytotoxic chemotherapy more than 30 days prior to entry.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Malabsorption or severe chronic diarrhea within 30 days prior to entry, or inability to consume adequate oral intake because of chronic nausea, emesis, or abdominal or esophageal discomfort.
* Inadequately controlled seizure disorder.
* Known intolerance to stavudine, didanosine, and/or hydroxyurea.
* Acute and clinically significant medical event within 30 days of screening.
* Any clinical or laboratory abnormality greater than Grade 3 toxicity, with the exception of laboratory values given.

Concurrent Treatment:

Excluded:

- Any experimental antiretroviral therapy or immunomodulators directed against HIV-1, e.g., IL-4, cyclosporine steroids at doses greater than 40 mg/day.

Prior Medication:

Excluded:

- Non-nucleoside reverse transcriptase inhibitor therapy.

Prior Treatment:

Excluded:

* Radiation therapy within 30 days of entry except to a local lesion.
* Transfusion of blood or blood products within 21 days of screening.
* Cytotoxic therapy within 3 months of study entry.

Risk Behavior:

Excluded:

Active substance abuse that may interfere with compliance or protocol evaluations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Dr Robert Wallace, St. Petersburg, Florida, United States